CLINICAL TRIAL: NCT06475300
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of BL-B01D1+PD-1 Monoclonal Antibody in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer, Nasopharyngeal Carcinoma and Other Solid Tumors
Brief Title: A Study of BL-B01D1+PD-1 Monoclonal Antibody in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer, Nasopharyngeal Carcinoma and Other Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-204-05
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer; Nasopharyngeal Carcinoma; Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Nasopharyngeal Carcinoma | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1+PD-1 Monoclonal Antibody (Experimental): Participants receive BL-B01D1+PD-1 Monoclonal Antibody as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: PD-1 Monoclonal Antibody

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: PD-1 Monoclonal Antibody — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This phase II study is a clinical study to explore the efficacy and safety of BL-B01D1 combined with PD-1 Monoclonal Antibody in patients with locally advanced or metastatic non-small cell lung cancer, nasopharyngeal carcinoma and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Any gender;
3. Age: ≥18 years old;
4. Expected survival time for 3 months or more;
5. Patients with locally advanced or metastatic non-small cell lung cancer or nasopharyngeal carcinoma confirmed by histopathology and/or cytology;
6. Subjects were able to provide 6-10 slides of archived tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 2 years;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. ECOG 0 or 1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No serious cardiac dysfunction, left ventricular ejection fraction 50% or higher;
11. screening period not allowed within 14 days before a blood transfusion, are not allowed to use any cell growth factor, and/or liters of platelet medicine, organ function level must conform to the requirements;
12. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5ULN;
13. The urine protein + 2 or 1000 mg / 24 h or less or less;
14. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, serum or urine must be negative for pregnancy, and must be non-lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Stage 1 EGFR-sensitive mutant non-small cell lung cancer patients with systemic chemotherapy; Stage 2 patients who had received previous systemic therapy;
2. In the second stage queue one signed informed consent before gene sequencing report suggests patients such as mutation of ALK fusion;
3. Anti-tumor therapy such as chemotherapy or biological therapy has been used within 4 weeks or 5 half-lives before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Fluorouracil class oral drugs, etc.;
4. Serious heart disease;
5. Long QT, complete left bundle branch block, III degree atrioventricular block; Serious arrhythmia;
6. Active autoimmune and inflammatory diseases;
7. Before the first delivery within 5 years diagnosed as other malignant tumor;
8. Two antihypertensive drugs poorly controlled hypertension;
9. Patients with poor glycemic control;
10. With a history of ILD, current ILD or suspected suffering from such diseases during screening;
11. Complicated with pulmonary diseases leading to severe respiratory function impairment;
12. There is a lot of serous cavity effusion, or have a serous cavity effusion and has symptoms, or poorly controlled serous cavity effusion patients;
13. Imaging studies suggest tumor has violated or package around the chest, neck, pharyngeal large blood vessels;
14. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
15. Active central nervous system of patients;
16. For restructuring or human mouse chimeric antibody on study of humanized anti-platelet antibody has a history of allergies or allergic to BL - B01D1 any supplementary material composition of patients;
17. Before transplant or allogeneic hematopoietic stem cell transplantation (Allo - HSCT);
18. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
19. Active infection requiring systemic therapy;
20. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
21. Had participated in another clinical trial within 4 weeks before the first dose;
22. Other conditions for trial participation were not considered appropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China